CLINICAL TRIAL: NCT06773117
Title: Efficacy/Safety of Susu Xiao'er Zhike Granules for Children's Cold-Induced Cough (Wind-Cold Syndrome): Multicenter, Randomized, Double-Blind, Low-Dose Controlled Phase III Trial
Brief Title: Phase III Trial of Susu Zhike Granules in Children With Cold-cough Syndrome for Acute Cough Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-SSXEZKKL-Ⅲ
Record Dates: First submitted 2024-08-30; First posted 2025-01-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Susu Xiao'er Zhike Granules 1 bag
  Interventions: Drug: Susu Xiao'er Zhike Granules
- control group (Other): Extremely-low dose Susu Xiao'er Zhike Granules 1 bag
  Interventions: Drug: Extremely-low dose Susu Xiao'er Zhike Granules

INTERVENTIONS:
Drug: Susu Xiao'er Zhike Granules — Susu Xiao'er Zhike Granules 1 bag(7g granule per bag,contains 20.25 g crude herbs), twice a day for five days
  Arms: experimental group
Drug: Extremely-low dose Susu Xiao'er Zhike Granules — Extremely-low dose Susu Xiao'er Zhike Granules 1 bag (7g granule per bag,contains 1.01 g crude herbs), twice a day for five days
  Arms: control group

SUMMARY:
To confirm the effect of Susu Xiaoer Zhike granules in treating cough caused by common cold (wind-cold cough Syndromes) in children aged 6~13 years, shortening the course of disease and improving symptoms.

DETAILED DESCRIPTION:
Susu used to be a clinical experienced Chinese herb formula for treating acute cough caused by common cold. The ingredients includes Hua Ju Hong, Qiao Rui Su, Zi Su Ye, Jie Geng, Gan Cao,which relieving cold and cough, resolving phlegm in traditional Chinese medicine theory. This prescription was used for a long time in clinical for treatingacute cough caused by common cold as an herb formula. To standardize the quality and make it easier to take, The investigators reproduced it into a patent medicine and design this trial for evaluating it.

The phase II clinical study of Susu Xiaoer Zhike Granules was carried out in the past, and the results showed that the use of Susu Xiaoer Zhike granules (containing 20.25g of raw drug) in the high dose group could significantly improve the clinical recovery rate (P<0.05) and shorten the clinical recovery time (P<0.05) in children aged 6 to 14 years (< 14 years) caused by common cold (wind-cold cough). And good security. Based on the effectiveness and safety results of the phase II clinical study, this study intends to select the high-dose group of the phase II clinical study (containing 20.25g of raw drug) as the experimental group of the phase III clinical study, and the extremely-low dose group of the phase II clinical study as the control group. To conduct confirmatory clinical studies on cough (wind-cold cough) caused by common cold in children aged 6 to 13 years (6 years ≤ age < 14 years).

ELIGIBILITY:
Inclusion Criteria:

1. It met the diagnostic criteria for common cold, and the severity VAS score of day or night cough was ≥40 mm ，the cough symptom score was ≥2 points;
2. Conforming to the standard of wind-cold cough differentiation;
3. Age 6-13 years old (6 years old ≤ age < 14 years old);
4. Duration of cough ≤48 hours;
5. Maximum axillary temperature ≤38℃ within 24 hours before diagnosis;
6. The informed consent process should be in accordance with the regulations, and the legal guardian or the subject child (≥8 years old) should sign the informed consent.

Exclusion Criteria:

1. accompanied by pharyngeal swelling pain, heat image is obvious;
2. White blood cell count, neutrophils absolute value, C-reactive protein, all exceeded the upper limit of 1.2 times the reference value, and the researchers considered the bacterial infection;
3. there have been complications (bacterial otitis media, sinusitis, suppurative tonsillitis, bronchitis, bronchopneumonia);
4. Patients with acute bronchitis and pneumonia cured less than 8 weeks;
5. People with a history of seasonal or perennial allergic rhinitis, chronic sinusitis, chronic otitis media, bronchial asthma, chronic cough or recurrent respiratory infections;
6. Other acute episodes of nasal diseases (vasomotor rhinitis, drug rhinitis, etc.), nasal foreign body, or foreign body inhalation, any anatomical respiratory abnormalities;
7. Patients with serious systemic diseases or mental disorders such as cardiovascular, brain, liver, kidney and hematopoietic system;
8. Those who had used Chinese and Western drugs and therapies that had influence on the effectiveness evaluation of the experimental drugs within 24 h before enrollment;
9. Allergic to known components of the investigational drug;
10. Those who participated in other clinical trials and took investigational drugs within the past one month;
11. Those who were not considered suitable for inclusion by the researchers.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cough disappearance rate | 5 days
  Cough symptom scores were recorded at baseline and daily after treatment and evaluated at the end of treatment (Patients whose cough did not disappear were followed up for 24 hours).

SECONDARY OUTCOMES:
Cough symptom score | Baseline, 1, 2, 3, 4, and 5 days
  Baseline and post-treatment were recorded daily, and diachronic changes were evaluated at the end of treatment.
VAS score of cough symptoms | Baseline, 1, 2, 3, 4, and 5 days
  Baseline and post-treatment were recorded daily, and diachronic changes were evaluated at the end of treatment.
Time to disappearance of cough | 5 days
  Cough symptom scores were recorded at baseline and daily after treatment and evaluated at the end of treatment (Patients whose cough did not disappear were followed up for 24 hours).
Onset time of cough | 5 days
  Cough VAS score were recorded at baseline and daily after treatment and evaluated at the end of treatment
Disease cure rate | 5 days
  Cold symptoms were recorded and evaluated at baseline and after 5 days of treatment.
PAC-QoL scale score | 5 days
  Baseline and 5 days of treatment were recorded and evaluated.
Effective rate of TCM syndrome | 5 days
  Baseline and 5 days of treatment were recorded and evaluated.
The rate of disappearance of individual symptoms | 5 days
  Baseline and 5 days of treatment were recorded and evaluated.
Incidence OF COMPLICATIONS | 5 days
  Post-treatment records were recorded and end-of-treatment evaluations were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Li, Study Chair — The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine
Locations (19):
- China (19):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Jiangjin District Central Hospital of Chongqing, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Zunyi First People's Hospital, Zunyi, Guizhou
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Zhengzhou First People's Hospital, Zhengzhou, Henan
  - Sinopharm Dongfeng General Hospital, Shiyan, Hubei
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changshang, Huna
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Wuxi Eighth People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Yanbian University (Yanbian Hospital), Yanji, Jilin
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - Changzhi People's Hospital, Changzhi, Shanxi
  - The Affiliated Hospital of Chengdu University of Chinese Medicine, Chengdu, Sichuan
  - The First Teaching Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality
  - Tianjin Children's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No